CLINICAL TRIAL: NCT01341587
Title: Comparison of a Cellular-embedded Glucose Meter With Two-way Personalized Communication Between Patients and Care Managers With a Glucose Meter in Standard Practice in the Care of Diabetic Patients.
Brief Title: Smart Glucose Meter Project
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: participants lost to follow-up;
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Maryland Industrial Partnerships (Other); Telcare, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00045527
Record Dates: First submitted 2011-02-07; First posted 2011-04-25 (Estimated); Results first posted 2018-03-12 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2019-12

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
Keywords: SMBG (self monitoring of blood glucose); diabetes; mobile technology
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Provider-driven care, based in office, no special diabetes management; Patient self-monitoring of blood glucose (SMBG)
- Intervention (Active Comparator): Home diabetes monitoring by patient using cellular enabled glucometer to communicate information and receive feedback.
  Care provider can access raw and analyzed patient data; Physician receives report summary.
  Interventions: Device: Telcare Blood Glucose Meter (BGM)

INTERVENTIONS:
Device: Telcare Blood Glucose Meter (BGM) — Cellular enabled glucometer
  Arms: Intervention

SUMMARY:
Currently, in the U.S., 1 in 3 males and 2 in 5 females born after 2000 are expected to develop diabetes during his or her lifetime. Research has demonstrated that control of blood glucose (BG) reduces the complications of diabetes. As a result, almost half of Americans diagnosed with diabetes, are prescribed finger-stick glucose meters to monitor their BG. The value of this approach is known to be limited by a high rate of patient non-compliance with BG testing, where patients test less often than prescribed. Increased communication between patient and care manager along with feedback has been shown to increase self monitoring of blood glucose (SMBG) test compliance. However, this feedback loop is largely absent from the current, episodic model of patient / care manager interaction and not available in existing BG meters given to diabetic patients.

In this study, we propose to pilot test a cellular-embedded glucose meter. This device can transmit glucose readings directly over a cellular network to a care management server and then the patient will receive feedback on the screen of the glucose meter.

DETAILED DESCRIPTION:
This research program will enroll participants in a 6-month pilot intervention study. In this study, 100 patients with diabetes (Type 1 and Type 2) who are known to be non-compliant with SMBG will be enrolled and randomized to treatment groups (one group will receive a standard glucose meter and the second group will receive the cellular-embedded device) in order to achieve the following specific study aims;

Primary Aim 1: Determine if connecting diabetic patients to care managers via a cellular-enabled glucose meter with feedback will improve SMBG testing compliance.

Secondary Aim 2: Determine if increased testing compliance leads to improvement in overall blood glucose control. This will be measured by a reduction of HbA1c levels.

Secondary Aim 3: Determine whether this intervention leads to significant improvements in patient satisfaction with self-care and patient self-assessment of compliance.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Diagnosis of Diabetes Mellitus (Type 1 or Type 2)
* Currently, non-compliant with prescribed glucose testing regimen
* HbA1c of 7.5 or greater within the last six months

Exclusion Criteria:

* Actively being treated for substance abuse
* Treatment for a thought disorder within the past year
* Non-English speaking
* Persons who are legally blind
* Women who are pregnant
* Cognitively or decisionally impaired as determined by practitioner
* Persons using an insulin pump

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Geppi, Study Director — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Home diabetes monitoring by patient using cellular enabled glucometer to communicate information and receive feedback.
  Care provider can access raw and analyzed patient data; Physician receives report summary.
  Telcare Blood Glucose Meter (BGM): Cellular enabled glucometer
Period: Overall Study
Arm/Group | Control | Intervention
Started | 4 | 10
Completed | 0 | 0
Not Completed | 4 | 10
Not completed — Lost to Follow-up | 2 | 0
Not completed — stopped using the meters | 2 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 4 | 10 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (18) | 52.8 (13.4) | 52.3 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 2 | 6 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 9 | 13
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 10 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c
Description: Determine whether this intervention leads to significant improvements in patient HbA1c from baseline to 6 months
Time Frame: 6 months
Population: Results for change were not collected because the study was stopped. Participants were lost to follow-up and stopped using the meters
Arm/Group | Control | Intervention
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Control | Intervention
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/10
Other Adverse Events (participants affected / at risk) | 0/4 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No